CLINICAL TRIAL: NCT03914807
Title: Cow Milk Fat Obesity pRevention Trial
Acronym: CoMFORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Jonathon L Maguire, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-369
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Obesity, Childhood
Keywords: milk; fat; cohort-embedded
MeSH Terms: conditions — Pediatric Obesity; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Intervention Model Description: Superiority cohort embedded 2 arm pragmatic randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole (3.25%) milk (Active Comparator)
  Interventions: Other: Whole (3.25%) cow's milk recommendation
- Reduced fat (1%) milk (Active Comparator)
  Interventions: Other: Reduced (1%) fat milk

INTERVENTIONS:
Other: Whole (3.25%) cow's milk recommendation — Children randomized to the whole milk recommendation will receive a recommendation a primary care recommendation to consume 500 mL of whole fat (3.25%) milk instead of transitioning to reduced fat (1%) milk at 2 years of age. The primary care physician will verbally make this recommendation during the recruitment well-child visit. Parents will also be reminded bi-monthly by phone calls made by a research assistant. Children in the whole milk recommendation group will be provided with the same age-appropriate nutritional recommendations as children in the reduced fat recommendation group as part of routine healthcare according to the Rourke Baby Record.
  Arms: Whole (3.25%) milk
Other: Reduced (1%) fat milk — Children randomized to the reduced fat group will receive a primary care recommendation to transition from whole milk to 500 mL reduced fat (1%) milk daily once the child is two years of age (consistent with current guidelines). The physician will verbally make this recommendation during the recruitment well-child visit. Parents will also be reminded bi-monthly by phone calls made by a research assistant. Children who receive the reduced fat recommendation will be provided with the same age-appropriate nutritional recommendations as children who receive the whole fat recommendation as part of routine healthcare according to the Rourke Baby Record.
  Arms: Reduced fat (1%) milk

SUMMARY:
Cow's milk is a dietary staple for children in North America. Though clinical guidelines suggest children transition from whole (3.25% fat) milk to reduced (1%) fat milk at age 2 years, recent epidemiological evidence supports a link between whole milk consumption and lower adiposity in children. The purpose of this trial is to determine which milk fat recommendation minimizes excess adiposity and optimizes child nutrition and development. CoMFORT will be a parallel group randomized controlled trial among children aged 2 to 4 years participating in the TARGet Kids! practice-based research network. Children will be randomized to receive one of two usual care nutritional recommendations: 1) a recommendation to consume whole milk, or 2) a recommendation to consume reduced (1%) fat milk. The primary outcome is Body Mass Index z-score (zBMI); secondary outcomes will be cognitive development (using the Ages and Stages Questionnaire), vitamin D stores (serum 25-hydroxyvitamin D), cardiometabolic health (glucose, hsCRP, non-HDL, LDL, triglyceride, HDL and total cholesterol, insulin, and diastolic and systolic blood pressure) and sugar sweetened beverage intake (measured by 24-hour dietary recall). Outcomes will be measured 24 months post-randomization and compared using ANCOVA, adjusting for baseline measures. This trial will contribute to nutrition policy for children in effort to reduce childhood obesity using a simple, inexpensive and scalable cow's milk fat intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy by parental report;
* 1.5 to 2.99 years of age
* involved in a TARGet Kids! academic pediatric or family medicine group.

Exclusion Criteria:

* Prader-Willi syndrome or other syndrome associated with obesity
* severe development delay
* children who are from families without verbal communication in English or French
* failure to thrive (with zBMI values ≤ -2 are unlikely to benefit from obesity prevention)
* siblings of trial participants as families may share milk
* will not consume cow's milk by choice, lactose intolerance or allergy.

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 534 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
weight | Measured 24 months post-study entry
  kilograms; measured using a Healthometer stadiometer
height | Measured 24 months post-study entry
  metres; measured using a Healthometer statiometer
body mass index z-score (zBMI) | Measured 24 months post-study entry
  BMI calculated by weight (kg)/height (m^2); zBMI determined according to the World Health Organization guidelines

SECONDARY OUTCOMES:
serum 25-hydroxyvitamin D | Measured 24 months post-study entry
  measured in nmol/L
serum glucose | measured 24 months post-study entry
  measured in mmol/L
blood pressure | measured 24 months post-study entry
  systolic and diastolic
serum insulin | measured 24 months post-study entry
  measured in mmol/L
serum triglycerides | measured 24 months post-study entry
  measured in mmol/L
serum total cholesterol | measured 24 months post-study entry
  measured in mmol/L
serum high density lipoprotein cholesterol | measured 24 months post-study entry
  measured in mmol/L
serum low density lipoprotein cholesterol | measured 24 months post-study entry
  measured in mmol/L
serum non-high density lipoprotein cholesterol | measured 24 months post-study entry
  measured in mmol/L
serum highly sensitive c-reactive protein | measured 24 months post-study entry
  measured in mg/L
height z-score | measured 24 months post-study entry
  measured by a trained research assistant according to the World Health Organization guidelines
waist circumference | measured 24 months post-study entry
  measured by a trained research assistant
lean body mass | measured 24 months post-study entry
  measured in kg, % body weight
fat mass | measured 24 months post-study entry
  measured in kg, % body weight
school readiness | measured 24 months post-study entry
  measured using the Early Development Instrument (EDI); children scoring at or below the 25th percentile of children in their province are considered at risk for continuing on the low achievement and health trajectory, and are more likely to fall behind in academic achievement in later grades
cognitive development | measured 24 months post-study entry
  measured using the Ages and Stages Questionnaire (ASQ)
dietary intake | measured 24 months post-study entry
  measured using the Automated Multiple Pass Self Administered 24 hour recall (ASA24) tool
carotid intima media thickness (cIMT) | measured 24 months post-study entry
  measured by ultrasound
restrained and emotional eating | measured 24 months post-study entry
  measured using the 3-factor eating questionnaire
nutritional risk | measured 24 months post-study entry
  measured using NutriSTEP preschooler
physical activity (minutes per day) | measured 24 months post-study entry
  questionnaire data and accelerometry
sleep time (hours per night) | measured 24 months post-study entry
  questionnaire data and accelerometry
healthcare service utilization | measured 24 months post-study entry
  information accessed through OHIP linkage
upper respiratory tract infection incidence | measured 24 months post-study entry
  information accessed through OHIP linkage
growth trajectories | measured 24 months post-study entry
  zBMI growth rates
head circumference | measured 24 months post-study entry
  measured by a trained research assistant
cost effectiveness | measured 24 months post-study entry
  All costs, parameter estimates and ranges will be derived from study data and will be obtained using medical record extraction. Publicly available Ontario costing sources will be used to cost resource utilisation parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon L Maguire, MD, FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanderhout SM, Aglipay M, Birken C, Li P, O'Connor DL, Thorpe K, Constantin E, Davis MA, Feldman M, Ball GDC, Janus M, Juni P, Junker A, Laupacis A, L'Abbe M, Manson H, Moretti ME, Persaud N, Omand JA, Relton C, Wong P, Yamashiro H, Tavares E, Weir S, Maguire JL. Cow's Milk Fat Obesity pRevention Trial (CoMFORT): a primary care embedded randomised controlled trial protocol to determine the effect of cow's milk fat on child adiposity. BMJ Open. 2020 May 7;10(5):e035241. doi: 10.1136/bmjopen-2019-035241. PMID 32385063